CLINICAL TRIAL: NCT03558568
Title: The Effect of Subthalamic Nucleus Deep Brain Stimulation on Facial Expressions in Parkinson's Disease.
Brief Title: The Effect of Deep Brain Stimulation on Facial Expressions.
Acronym: STN-DBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Atilla YILMAZ, Assistant Professor, Mustafa Kemal University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1
Record Dates: First submitted 2018-05-28; First posted 2018-06-15 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Parkinson
Keywords: Parkinson's Disease; Deep Brain Stimulation; Subthalamic Nucleus; DBS; STN; Face; Facial expressions; Parkinson
MeSH Terms: conditions — Parkinson Disease; Facies; Facial Expression | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: The study initially recruited 18 patients with idiopathic PD who underwent DBS surgery for movement disorders caused by PD at Mustafa Kemal University Medical Faculty Neurosurgery Department.
  Inclusion criteria:
  * Idiopathic PD responsive to L-Dopa treatment,
  * Between 40-75 years of age,
  * Having received bilateral STN DBS surgery at least six months prior to the investigation to ensure stable stimulation parameters,
  * Mentally normal patients that could understand and respond to a directives.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- DBS off (Active Comparator)
  Interventions: Device: Deep Brain Stimulation
- DBS on 60 Hz. (Active Comparator)
  Interventions: Device: Deep Brain Stimulation
- DBS on 99 Hz. (Active Comparator)
  Interventions: Device: Deep Brain Stimulation
- DBS on 130 Hz. (Active Comparator)
  Interventions: Device: Deep Brain Stimulation
- DBS on 230 Hz. (Active Comparator)
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation is an established surgical method for Parkinson's Disease.
  Other Names: Vercise; Activa PC

SUMMARY:
Whether Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS), a treatment commonly used to ameliorate the motor symptoms of Parkinson's disease (PD), affects on facial expressions is unclear. The purpose of this study was to investigate the potential effects of DBS and different frequencies on facial expressions of PD patients by volunteers via a web site: http://www.supporttoscience.com

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most frequent progressive neuro-degenerative disease with a worldwide prevalence of 4-6 million and the mask face is an important and also troublesome sign of PD. Deep Brain Stimulation (DBS) surgery can be a viable option which has recently emerged and been accepted as a useful surgical method for PD. Standard DBS targets include Subthalamic Nucleus (STN) and Globus Pallidus Internus (GPi). Although the STN-DBS application is known to have favorable effects on motor and non-motor symptoms of PD, there is a lack information about the effect on facial expressions of PD patients. Our aim is to analyze the effect of the STN-DBS stimulation and different frequencies on the facial expressions of PD patients.

The study initially recruited 18 patients with idiopathic PD who underwent DBS surgery for movement disorders caused by PD at Mustafa Kemal University Medical Faculty Neurosurgery Department.

Inclusion criteria:

* Idiopathic PD responsive to L-Dopa treatment,
* Between 40-75 years of age,
* Having received bilateral STN DBS surgery at least six months prior to the investigation to ensure stable stimulation parameters,
* Mentally normal patients that could understand and respond to a directives. The evaluation will be made by the face photos of the patients. The face photos for the expressions including [normal], [sad], [happy], and [angry] were obtained at frequencies including 130 Hz, 60 Hz, 99 Hz, 230 Hz and off-stimulation. The face photos will evaluate by the software and by the volunteers with the aim of a website: http://www.supporttoscience.com

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD responsive to L-Dopa treatment,
* Between 40-75 years of age,
* Having received bilateral STN DBS surgery at least one month prior to the investigation to ensure stable stimulation parameters,
* Mentally normal patients that could understand and respond to a questionnaire.

Exclusion Criteria:

* Above 75 years of age,
* Severe dementia,
* History of an additional neurologic disease,
* The presence of a disease, such as the facial paralysis, that could affect facial expressions,
* Having a wound on the face.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-08-12 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
The effect of Deep brain stimulation on facial expressions will be analyzed by volunteers via a web site then the results will evaluate by statistical analyses. | 3 months
  The evaluation of patients photos (in different frequencies and when stimulation off status) will be analyzed by volunteers via a website, then the results will be compare and evaluate by statistical analysis. The results will give us an opinion about these:
  The effect of Deep Brain Stimulation on Parkinsonians patients facial expression and which frequency setting is better for facial expression.

CONTACTS AND LOCATIONS:
Locations (1):
- Atilla YILMAZ, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The results will be shared
URL: http://www.supporttoscience.com